CLINICAL TRIAL: NCT04935060
Title: The Acceptability and Feasibility of a Guide for Sharing the Outcome of a Memory Assessment
Brief Title: Sharing the Outcome of a Memory Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Northamptonshire Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20077
Record Dates: First submitted 2021-05-14; First posted 2021-06-22 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Dementia assessment (Active Comparator): Clinicians will conduct the assessment and outcome process as per their usual practice.
  Interventions: Behavioral: Usual Care
- Guide informed dementia assessment (Experimental): The guide will be used by both clinicians, patients and their companions to inform the approach to the dementia assessment process.
  Interventions: Behavioral: A guide to inform the process of delivering the outcomes of a dementia assessment

INTERVENTIONS:
Behavioral: A guide to inform the process of delivering the outcomes of a dementia assessment — The guide provides information that informs the approach taken to assessing people for dementia. It aims to guide clinicians. patients and their companions to think about how the diagnostic process is carried out, taking into account patient preferences, particularly around how they would like diagnostic decisions to be communicated to them.
  Arms: Guide informed dementia assessment
Behavioral: Usual Care — Clinicians conduct the dementia assessment as per standard protocols
  Arms: Usual Care Dementia assessment

SUMMARY:
The purpose of this study is to establish the acceptability of a guide developed to improve people's experiences of dementia assessment outcome appointments in comparison to a standard consultation. This study will also inform the feasibility of future research evaluating the guide and provide information on how well the measurements used provide evaluation of the intervention.

DETAILED DESCRIPTION:
Objectives:

To determine the acceptability of a guide supported consultation (intervention) for clinicians, patients and companions, in comparison to a standard diagnostic consultation (usual care).

To inform the feasibility of future research establishing recruitment processes and study uptake.

To establish how well the chosen measurement strategy provides evaluation of the intervention (including completion rates, perceived relevance and burdensomeness).

Setting:

NHS Secondary care, Memory Assessment Service (MAS). Services within the identified area are split into four teams. One team will provide the usual care treatment arm. Another team will provide the intervention arm.

Number of participants:

24 Patients and 24 Companions will be recruited for the quantitative component of the study.

Two clinicians and six participants will be recruited for the qualitative component of the study.

Description of interventions:

Baseline Measurement The Consultation and Relational Empathy (CARE) questionnaire and the adapted CARE (for companions) will be used to collect baseline data for each of the two sites. Baseline data will be collected from anyone attending outcome appointments at both sites during a recruitment period prior to the implementation of the intervention and will form an initial baseline cohort.

Quantitative Data Collection Usual Care Procedure The usual care procedure involves assessment of patient's cognitive abilities, daily functioning and physical health to determine the possibility of them having a dementia. This is done through a detailed history taking by MAS clinicians including information given by the patient, companions and information included from a GP referral. Standardised assessments are also conducted to inform the assessment process. These assessments are used based on the needs of the patient and companions involved. Access to scores on these assessments will be gained through their medical records and will provide a measurement for comparison between the two groups.

MAS outcome appointments are provided as part of routine care. These appointments require clinicians to rely on their professional judgement of the best way for the outcomes of assessments to be communicated to patients and their companions. There are no current standardised guidelines used within the service for this purpose.

In addition to the service's usual practice, participants will be asked to complete the CARE and the adapted CARE following their initial assessment and their outcome appointment. The completed questionnaires will be returned to the researcher by post via pre-paid envelope. A reminder via telephone call will be given to participants on the day following their appointment and if they haven't completed the questionnaire they will be given the opportunity to complete it whilst on the call with the researcher.

Intervention Procedure The intervention procedure will follow the same steps as the usual care procedure with the addition of use of the Bennett, De Boos and Moghaddam (2018) guide for clinicians, patients and companions. After gaining of written consent at the initial assessment appointment, the clinician will give the patient a copy of the guide and inform them that they can share this with their companion should they wish to. When conducting outcome appointments clinicians will use the guide to inform communication with the patient and companion. Clinicians will also refer patients and companions to their copy of the guide during the outcome appointment.

Qualitative Data Collection Qualitative data will be collected using semi-structured interviews with patients and companions as well as clinicians focussing on their experiences of the outcome appointment. Individuals taking part in the interviews will be involved will therefore be involved with the study for a further four weeks.

Duration of study:

Overall: March 2021-February 2022 Participants and companions involvement with the study will be for the duration of their assessment by the MAS teams. This is usually around 16 weeks but varies depending on the clinical needs of the patient. Participants taking part in the additional qualitative interview will extend the duration of their involvement in the study by up to four weeks.

Statistical Methods Quantitative data analysis Quantitative analysis will be descriptive and will aim to give confidence interval estimation. Baseline measures will be collected for each location to allow estimates of the variability between the two sites for comparison.

Intra Class Correlations (ICCs) will be carried out to examine the degree of clustering. Intention to treat (ITT) analysis will be carried out to give a more accurate estimate of effectiveness in clinical practice. Participants data will be analysed based on their experimental arm allocation.

Intra Class Correlations (ICCs) will be carried out to examine the degree of clustering. Intention to treat (ITT) analysis will be carried out to give a more accurate estimate of effectiveness in clinical practice. Participants data will be analysed based on their experimental arm allocation.

Viability of recruitment will be assessed using eligibility and consent rates for patients and clinicians. The burden of measure completion will be assessed through missing data levels as well as interviews with patients and clinicians. Withdrawal rates post consent will be calculated by study arm for use in future sample size calculations.

Qualitative data analysis A framework method, as set out by Ritchie and Spencer (1994), will be used to identify themes. This will allow for comparison of the experiences of participants in the two arms of the study. Analysis will follow the steps set out by Ritche and Spencer (1994); familiarisation, identifying a thematic framework, indexing, charting and mapping and interpretation.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if they are:

* Taking part in an initial assessment appointment with the participating MAS services
* Aged 18 years or over (Northamptonshire MAS require patients to be 65 years or over to be eligible for referral. There will be no upper age limit)
* Able to provide written informed consent

Companions will be included in the study if they are:

* Supporting a patient-participant to attend a MAS initial assessment appointment
* Aged 18 years or over
* Able to provide written, informed consent

MAS Clinicians will be included in the study if they are:

* Involved in the delivery of MAS outcome appointments
* Able to provide written informed consent

Exclusion Criteria:

* Patients and companions will not be included in the research if there is reason to doubt their capacity to give informed consent under the Mental Capacity Act 2005.
* Patients and companions who are not fluent in English will not be included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Difference in scores on The Consultation and Relational Empathy (CARE) Questionnaire for each condition | Baseline
  Measures patient and companions rating of clinician empathy in consultations. Higher scores suggest higher levels of clinician empathy. The maximum score possible is 50 and the minimum is 10.
Difference in scores on The Consultation and Relational Empathy (CARE) Questionnaire for each condition | Post initial Consultation. Up to four weeks following consultation appointment.
  Measures patient and companions rating of clinician empathy in consultations. Higher scores suggest higher levels of clinician empathy. The maximum score possible is 50 and the minimum is 10.
Difference in scores on The Consultation and Relational Empathy (CARE) Questionnaire for each condition | Post outcome appointment. Up to four weeks following outcome appointment.
  Measures patient and companions rating of clinician empathy in consultations. Higher scores suggest higher levels of clinician empathy. The maximum score possible is 50 and the minimum is 10.
Qualitative semi-structured interviews with patients and companions. | Interviews to take place following the outcome appointment. Up to four weeks following outcome appointment.
  Focussing on their experiences of the outcome appointment.
Qualitative semi-structured interviews with clinicians. | Interviews to take place within four weeks of clilnicians completing outcome appointments with all of the patients participating in the study.
  Focussing on their experiences of using the guide and delivering outcome appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle De Boos, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Memory Assessment Service (Corby/Kettering), Corby, Northamptonshire
  - Memory Assessment Service (Rushden/Wellingborough), Rushden, Northamptonshire

IPD SHARING:
Plan to Share IPD: No